CLINICAL TRIAL: NCT04298879
Title: A Phase 2, Multicenter, Open-Label Study of IBI376, a PI3Kδ Inhibitor, in Patients With Relapsed or Refractory Follicular Lymphoma/Marginal Zone Lymphoma
Brief Title: IBI376 in Patients With Relapsed or Refractory Follicular Lymphoma/Marginal Zone Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI376A201
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Indolent Non-hodgkin Lymphoma
Keywords: Follicular Lymphoma; Marginal Zone Lymphoma; Parsaclisib
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI376 (Experimental): IBI376 will be administered orally at a dose of 20 mg once daily for 8 weeks followed by 2.5 mg once daily.
  Interventions: Drug: IBI376

INTERVENTIONS:
Drug: IBI376 — IBI376 20 mg po. once daily for 8 weeks ，followed by 2.5mg once daily
  Other Names: Parsaclisib

SUMMARY:
A Phase 2, Multicenter, Open-Label Study of IBI376, a PI3Kδ Inhibitor, in Patients with Relapsed or Refractory Follicular Lymphoma/Marginal Zone Lymphoma

DETAILED DESCRIPTION:
Patients will be recruited for 2 cohorts. Cohort A will recruit 58 RRFL subjects, and Cohort B will recruit 62 RRMZL subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Histologically confirmed, relapsed or refractory, follicular B-cell non-Hodgkin lymphoma (NHL) (FL) Grade 1, 2, and 3a or MZL.
3. Ineligible for hematopoietic stem cell transplant.
4. Definition of RRFL or RRMZL: Subjects should have received 2 or more prior therapies for FL/MZL included at least one regimen containing Rituximab. Subjects should be refractory to Rituximab or experienced disease progression after achieved remission or disease progression within 6 months since last therapy.
5. Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of ≥ 1 lesion that measures > 1.5 cm in the longest dimension and ≥ 1.0 cm in the longest perpendicular dimension as assessed by computed tomography (CT) or magnetic resonance imaging (MRI).
6. Subjects must be willing to undergo an incisional, excisional, or core needle lymph node or tissue biopsy or provide a lymph node or tissue biopsy from the most recent available archival tissue.
7. ECOG performance status 0 to 2.
8. Life expectancy ≥ 12 weeks.
9. Adequate hematologic, hepatic, and renal function.
10. Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

1 . Known histological transformation from indolent NHL to diffuse large B-cell lymphoma.

2. History of central nervous system lymphoma (either primary or metastatic).

3. Prior treatment with idelalisib, other selective PI3Kδ inhibitors, or a pan-PI3K inhibitor.

4. Prior treatment with a Bruton's tyrosine kinase inhibitor (eg, ibrutinib).

5. Allogeneic stem cell transplant within the last 6 months, or autologous stem cell transplant within the last 3 months before the date of study treatment administration.

6. Active graft-versus-host disease. 7. Subjects positive for hepatitis B surface antigen or hepatitis B core antibody will be eligible if they are negative for HBV-DNA. Subjects positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  To assess the efficacy of IBI376 in terms of objective response rate (ORR) in subjects with relapsed or refractory follicular lymphoma (FL)/Marginal lymphoma(MZL). Subjects will be evaluated for ORR by an IRC (Lugano criteria)

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | 2 years
  To assess complete response rate (CRR)
Duration of Response (DOR) | 2 years
  To assess the duration of response (DOR)
Progression-free Survival (PFS) | 2 years
  To assess progression-free survival (PFS)
Overall Survival (OS) | 2 years
  To assess overall survival (OS)
Best percentage change in target lesion size | 2 years
  To assess best percentage change in target lesion size
Safety and tolerability of IBI376 measured by adverse events (AEs) | Baseline through 30-35 days after end of treatment, up to approximately 12 months per subject
  Defined as any AE either reported for the first time or worsening of a pre-existing event after first dose of study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, school of medicine, Shanghai jiao tong university, Shanghai, China